CLINICAL TRIAL: NCT01453543
Title: The Effect of Deep Friction Massage on the Achilles Tendon Blood Flow
Acronym: Friction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/460
Record Dates: First submitted 2011-10-12; First posted 2011-10-18 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Healthy Situation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deep transverse friction massage (Experimental): Massage technique will be used.
  Interventions: Other: deep transverse friction massage

INTERVENTIONS:
Other: deep transverse friction massage — For the application of the deep transverse friction massage, the participants were positioned supine with the ankle in 90 ° of dorsiflexion, in order to bring some tension on the tendon. The treating clinician stabilized the subject's foot with one hand while applying the DTF with the other hand. The deep friction massage is a pinching technique with thumb and index finger, reinforced by the middle finger.

SUMMARY:
Background: There is a hypothesis in literature that the mechanical action of deep transverse friction massage (DTF) produces vasodilatation and increases blood flow. But as yet, no experimental study has confirmed the effect of DTF on blood flow in the Achilles tendon. Objective: The purpose of the present study was to investigate whether one session of DTF can influence the Achilles tendon blood flow.

Design: a randomized pre- posttest trial was set up. Patients: Sixty-two healthy participants volunteered. Each person underwent the following four steps of the procedure: 1. Measuring the tendon blood flow (PRE), 2.fifteen minutes of DTF on the Achilles tendon, 3. Measuring of the tendon blood flow (POST), 4.follow - up measurement after 20 minutes of rest (POST20).

Intervention: one leg of each person was randomly assigned to deep transverse friction session, the other leg was used as a control leg. Friction was applied continuously for a total of 15 minutes. Measurements: the microcirculation was determined at 2 and 8 tissue depths at the distal and the proximal midportion of the Achilles tendon. For each level, the capillary blood flow, the tissue oxygen saturation, and the postcapillary venous filling pressure was registered.

ELIGIBILITY:
Exclusion Criteria:

* a history of lower leg injury
* systematic disease
* persons using drugs
* subjects with circulatory disorders or cardiovascular diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Blood flow of the Achilles tendon | after 15 minutes of friction
  Blood flow of the Achilles tendon will be measured with the oxygen-to-see.
Blood flow of the Achilles tendon | After 20 minutes of rest.
  Blood flow of the Achilles tendon will be measured with the oxygen-to-see.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Witvrouw, MD, PhD, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium